CLINICAL TRIAL: NCT06843486
Title: Strong Bones: Promoting Bone Health and Quality of Life in Postmenopausal Women.
Brief Title: SB: Promoting Bone Health in Women
Acronym: SB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Politécnico de Bragança (Other)
Responsible Party: Principal Investigator, André Schneider, Principal Investigator, Instituto Politécnico de Bragança
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 755614
Record Dates: First submitted 2025-02-05; First posted 2025-02-25 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Womens; Menopause
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): The group will not receive any type of intervention
- Multicomponent Exercise (Experimental): Participants receive an intervention (a multi-component exercise program).
  Interventions: Other: Multicomponent Exercise

INTERVENTIONS:
Other: Multicomponent Exercise — Training sessions will include aerobic, resistance, balance and flexibility exercises, following the American College of Sports Medicine (ACSM) guidelines for osteoporosis prevention.
  Arms: Multicomponent Exercise

SUMMARY:
The goal of this clinical trial is to find out whether multicomponent training works to treat osteoporosis in women. It will also find out about the safety of multicomponent training in this specific population. The main questions it aims to answer are:

Does multicomponent training improve bone mineral density in women?

What are the benefits of multicomponent training?

The researchers will compare the intervention group (MTC) with a control group that did not perform any type of intervention, to see if MTC training works in treating bone mineral density in women.

The participants will:

Perform MTC training for 6 months with a frequency of 3 times a week in sessions of 40-60 minutes. While the control group will carry out their daily activities normally and will only attend on the days of the assessments.

DETAILED DESCRIPTION:
The Strong Bones Project is a randomized controlled trial (RCT) investigating the effects of Multicomponent Training (MCT) on bone mineral density (BMD), quality of life, and risk of osteoporosis in women.

The study adopts a hybrid approach combining cross-sectional observational analyses and randomized experimental interventions. Participants will be randomly allocated to an intervention group and a control group, allowing comparison of the impacts of MCT.

The interventions include a structured physical exercise program, with three distinct approaches:

1. In-Person Supervised Multicomponent Training (MCT In-Person)
2. Control Group (No active intervention, only clinical monitoring)

Training sessions will include aerobic, resistance, balance, and flexibility exercises, following the American College of Sports Medicine (ACSM) guidelines for osteoporosis prevention.

Data collection will include:

* Sociodemographic data
* Bone mineral density (BMD), assessed by DXA (Dual-Energy X-ray Absorptiometry)
* Functional fitness tests (e.g. handgrip strength test)

Participants will be followed for 6 months, with monthly assessments to monitor the progression of clinical variables.

Expected results include improved bone density, reduced risk of fractures, and improved quality of life.

The findings will be disseminated through scientific publications in peer-reviewed journals and presentations at international conferences on bone health and physical exercise.

This study seeks to contribute to the formulation of personalized physical exercise guidelines for the prevention of osteoporosis, especially in premenopausal women and men at intermediate risk of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Women over 65 years of age. Clinical diagnosis:

Previous diagnosis of osteoporosis confirmed by DXA (T-score between -1.0 and -2.5 for osteopenia and ≤ -2.5 for osteoporosis).

* Ability to exercise: Medical clearance to participate in the exercise program. and ability to perform moderate-impact physical activities and muscular endurance.
* Level of physical activity: Sedentary women or women with low to moderate levels of physical activity, without regular practice of specific exercises for bone health in the last 6 months.
* Agreement to the study: Signing of the Free and Informed Consent Form (FICF) and availability to participate in the training program for 6 months.

Exclusion Criteria:

* Advanced clinical diagnosis: T-score below -3.0 (severe osteoporosis with high risk of fractures); History of severe osteoporotic fracture in the last 6 months.
* Associated diseases or conditions: Uncontrolled metabolic or endocrine diseases that affect bone metabolism (e.g., hyperparathyroidism, Cushing's syndrome, decompensated diabetes); Active chronic inflammatory diseases (e.g., advanced rheumatoid arthritis, systemic lupus erythematosus); Severe chronic renal failure (stages 4 or 5).
* Use of specific medications in the last 12 months: Bisphosphonates, denosumab, teriparatide or strontium ranelate; High-dose glucocorticoids (>5 mg/day for more than 3 months); Recent hormone therapy for osteoporosis.
* Orthopedic or neuromuscular conditions: Severe functional limitation that prevents the performance of physical exercises (e.g., severe osteoarthritis, advanced joint instability, neurological sequelae of stroke); Orthopedic surgery in the last 6 months or indication for elective surgery for the spine or lower limbs.
* Factors that limit adherence to the study: Difficulty in moving that prevents participation in in-person training (for the in-person MCT group); Lack of availability to attend sessions or follow the study protocol; History of low adherence to previous health-related interventions.
* Participation in another clinical study: Women enrolled in clinical trials that may interfere with the results of the study or adherence to the protocol.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (BMD) | From enrollment to the end of treatment at 6 months
  Bone mineral density (BMD), measured in g/cm², assesses regions such as the lumbar spine, proximal femur, and total body. It is used to diagnose and monitor osteopenia and osteoporosis based on WHO criteria. The T-score, expressed in standard deviations (SD), compares the patient's BMD to that of a young, healthy population, classifying osteopenia (T-score -1.0 to -2.5 SD) and osteoporosis (T-score ≤ -2.5 SD). The Z-score compares BMD to age- and sex-matched averages, aiding in identifying secondary causes of osteoporosis.
  Dual-energy X-ray absorptiometry (DXA) is the standard method for measuring BMD. Additionally, DXA provides body composition analysis, offering data on bone mass (grams), lean mass (grams/kilograms), and body fat percentage (%). These parameters enable a comprehensive assessment of musculoskeletal health and nutritional status.

SECONDARY OUTCOMES:
Lower Limb Strength | From enrollment to the end of treatment at 6 months
  Test: 30-Second Chair Stand Description: Participants sit on a standard chair (43 cm height) and stand up as many times as possible within 30 seconds, without using their arms for support.
  Unit of Measure: Number of repetitions in 30 seconds
Upper Limb Strength | From enrollment to the end of treatment at 6 months
  Test: Arm Curl Test Description: Participants perform as many full biceps curls as possible within 30 seconds while holding a dumbbell (2.27 kg for women).
  Unit of Measure: Number of repetitions in 30 seconds
Lower Limb Flexibility | From enrollment to the end of treatment at 6 months
  Test: Chair Sit-and-Reach Test Description: Participants sit on the edge of a chair with one leg extended and reach toward their toes.
  Unit of Measure: Distance between fingers and toes (centimeters)
Upper Limb Flexibility | From enrollment to the end of treatment at 6 months
  Test: Back Scratch Test Description: Participants attempt to touch their fingertips behind their back, reaching one arm over the shoulder and the other behind the back.
  Unit of Measure: Distance between middle fingers (centimeters)
Agility/Balance | From enrollment to the end of treatment at 6 months
  Test: Timed Up and Go (TUG) Test Description: Participants stand up from a chair, walk 2.45 meters, turn around, and return to the seated position as quickly as possible.
  Unit of Measure: Time to complete the test (seconds)
Aerobic Endurance | From enrollment to the end of treatment at 6 months
  Test: 2-Minute Step Test Description: Participants march in place for two minutes, ensuring that their knee reaches a predefined height (midpoint between patella and iliac crest).
  Unit of Measure: Number of times the right knee reaches the marked height

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Politécnico de Bragança, Bragança, Braganza District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR